CLINICAL TRIAL: NCT06085313
Title: Cancer Pain Management: A Technology-Based Intervention for Asian American Breast Cancer Survivors
Brief Title: Cancer Pain Management Using a Web-based Intervention
Acronym: CAI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00004807
Record Dates: First submitted 2023-10-02; First posted 2023-10-16 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Cancer of Breast; Depressive Symptoms; Cancer Pain
MeSH Terms: conditions — Breast Neoplasms; Depression; Cancer Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAI: Web App-based, individualized coaching and support program for cancer pain (Experimental): Web App-based information and coaching/support program for cancer pain management with the individual optimization functionality
  Interventions: Behavioral: CAI
- CAPA: Web App-based information and coaching/support program for cancer pain (Active Comparator): Web App-based information and coaching/support program for cancer pain management
  Interventions: Behavioral: CAPA

INTERVENTIONS:
Behavioral: CAI — Web App-based information and coaching/support program for cancer pain management with additional components for the individual optimization functionality
  Arms: CAI: Web App-based, individualized coaching and support program for cancer pain
Behavioral: CAPA — Web App-based information and coaching/support program for cancer pain management
  Arms: CAPA: Web App-based information and coaching/support program for cancer pain

SUMMARY:
This study is funded by the HEAL Initiative (https://heal.nih.gov/). Based on Preliminary Studies (PSs), the research team developed and pilot-tested an evidence-based Web App-based information and coaching/support program for cancer pain management (CAPA) that was culturally tailored to Asian American breast cancer survivors using multiple unique features. However, CAPA rarely considered depressive symptoms accompanying pain in its design or components, and PSs indicated the necessity of further individualization of the intervention components of CAPA due to diversities in the needs of ABD. The purpose of the proposed 2-phase study is to further develop CAPA with additional components for ABD and the individual optimization functionality (CAI) and to test the efficacy of CAI in improving cancer pain experience of ABD. The specific aims are to: a) develop and evaluate CAI through an expert review and a usability test (R61 phase); b) determine whether the intervention group (that uses CAI and usual care) will show significantly greater improvements than the active control group (that uses CAPA and usual care) in primary outcomes (cancer pain management and cancer pain experience including depressive symptoms) from baseline to post 1-month and post 3-months; c) identify theory-based variables (attitudes, self-efficacy, perceived barriers, and social influences) that mediate the intervention effects of CAI on the primary outcomes; and d) determine whether the effects of CAI on the primary outcomes are moderated by selected background, disease, genetic, and situational factors. This study is guided by the Bandura's Theory and the stress and coping framework by Lazarus and Folkman. The R61 phase includes: (a) the intervention development process, (b) a usability test among 15 ABD, 15 family members, and 15 community gatekeepers; and (c) an expert review among 10 experts in oncology. The R33 phase adopts a randomized repeated measures control group design among 300 ABD. Long-term goals are: (a) to extend and test CAI in various healthcare settings with diverse subgroups of ABD, (b) examine the costeffectiveness, sustainability, and scalability of CAI in the settings, and (c) translate CAI into health care for ABD.

DETAILED DESCRIPTION:
Due to advances in early detection and treatment, breast cancer survivors represent nearly 70% of the 5.6 million female cancer survivors in the U.S. These women usually have some combination of surgery, radiation or chemotherapy, which can result in significant chronic pain. Indeed, the prevalence of pain is much higher in breast cancer survivors compared to survivors of other kinds of cancer. Pain occurs in 25%~60% of breast cancer survivors and about half report moderate to severe pain. Chronic pain decreases survivors' quality of life and daily functioning, and increases their fatigue, depression, anxiety, and sleep disruption.

Racial/ethnic minorities are high-risk groups for inadequate pain management. Racial/ethnic minority patients in the U.S. tend to present with a later-stage disease than non-minority patients, and their pain is more likely to be undertreated. Specifically, Asian Americans reportedly shoulder unnecessary burden of pain because they rarely complain, delay seeking help, and rarely ask necessary information or support due to cultural values, beliefs, and language barriers. Because of their cultural stigma attached to breast cancer, fear of addiction to pain medication, and stoicism toward pain, they tend to unnecessarily tolerate pain that they could easily manage with currently existing regimen including pharmacologic and non-pharmacologic strategies.

Especially, Asian American breast cancer survivors with depressive symptoms (ABD) are more likely to suffer from inadequate pain management due to their depression (e.g., not motivated enough to seek for help, stigma attached to depression), and pain could also worsen their depressive symptoms. Indeed, depression is a common co-morbidity in breast cancer survivors. A systematic literature review indicated that Asian American breast cancer survivors had moderate to high levels of depressive symptoms, anxiety and post-traumatic stress symptoms. In another study among 1,400 Chinese breast cancer survivors, about 26% had mild to severe depression and 13% fulfilled the criteria of clinical depression. Furthermore, as mentioned above, the recent opioid crisis has exacerbated their fear of addiction and reluctance to seek help. The Coronavirus Disease 2019 (COVID19) pandemic with Anti-Asian incidents has also placed an additional dimension of stress to this population.

Despite systematic efforts to provide adequate cancer pain management, researchers continue to find barriers including patients' beliefs and misconceptions, meanings of cancer pain, expectations about pain relief, miscommunication, lack of social support, inadequate training of healthcare providers and deficiencies within the healthcare infrastructure (e.g., insurance coverage). Among these, this study focuses on those at the individual and interpersonal levels of influence (by the National Institute of Minority Health and Health Disparity (NIMHD) Research Framework) as the first step.

Technology-based programs could be a solution to fill this gap in care for the survivors in communities. Mainly because of easy access (e.g., no transportation required, 24-hour access) and low cost (once the system is developed), technology-based programs are more effective in providing information and coaching/support than conventional program. Researchers also indicated their effectiveness in approaching isolated/ marginalized people with stigmatized conditions and underserved populations in communities. These marginalized groups report greater interest in e-health than their more affluent counterparts. In Preliminary Studies (PSs), Asian Americans preferred technology-based programs to traditional programs due to its high accessibility and anonymity. Furthermore, Internet use by Asian Americans is greater than that of any other racial/ethnic group, and over 93% of women are internet users.

Despite the strengths of technology-based programs, few technology-based interventions are available for breast cancer survivors, especially in pain and depressive symptom management. Little is known about the efficacy of culturally tailored technology-based interventions in improving pain and symptom experience of racial/ethnic minority cancer survivors, especially ABD. Only eight programs were identified in an extensive literature review. Two targeted individuals. One program had four face-to-face group sessions. Two programs combined face-to-face meetings with individual telephone counseling. One used a telephone conference approach. Two programs came from our own research team: one aimed to enhance general breast cancer survivorship experience (e.g., needs for help) by providing Web-based information and coaching/support (TICAA), and the other was CAPA that is the basis for CAI. CAPA has multiple unique features based on the actual data from PSs, which are rarely incorporated into technology-based interventions. Also, CAPA is the only existing technology-based program for cancer pain management that is culturally tailored to Asian American breast cancer survivors. However, CAPA rarely considers depressive symptoms accompanying pain in its design or components, and PSs indicated the necessity of further individualization of its components due to diversities in the needs of ABD. For instance, individual ABD selectively used only the specific online educational modules and resources that they were interested in.

CAI will offer the following features that have rarely been used in existing programs. First, CAI incorporates survivors' own cultural attitudes (deep tailoring) based on the actual data from PSs and uses multiple languages (surface tailoring). Indeed, cultural tailoring is essential in providing information and coaching/support for ABD because of their unique cultural heritage (e.g., Confucianism, stigma attached to breast cancer and depression, stoicism to pain). The use of multiple languages is also essential in providing information and coaching/ support to ABD who may not otherwise understand the material and instructions they are given. The feedback from community gatekeepers and ABD will be continuously incorporated into CAI as a part of the continuous cultural tailoring process. The impact of deep and surface tailoring will be differentiated in the dose-response analysis process (see Fidelity).

Second, the individual optimization functionality that will be developed in R61 Phase is unique because it allows further individualization of the intervention components for individual users through a machine-learning method (Genetic Algorithm). Through this functionality, CAI can deliver the most relevant and effective information and coaching/support to each participant. Because there exist diversities in ABD's needs for pain and depressive symptom management even within the same sub-ethnic group, this individualization is necessary; in PSs, ABD selectively used only those components that they were interested in.

Third, CAI is unique in incorporating both group (interpersonal level of influence) and individual (individual level of influence) coaching/support by culturally matched bilingual healthcare providers. There exist added benefits to protocols that include both group and individual coaching/support. Culturally matched bilingual interventionists could also ensure efficacy in coaching/support, limit the potential for harmful communications, provide reliable and objective information/resources, moderate and monitor liability or risk management issues, and nurture a positive group culture in culturally appropriate and sensitive ways.

Fourth, peer support through a social media function (interpersonal level of influence) is rarely used in existing programs. While social media as a health tool is understudied, findings indicate its effectiveness in providing information and coaching/support to breast cancer survivors including racial/ethnic minorities.

Finally, few existing programs incorporated existing evidence-based educational content from scientific authorities. Yet, the accuracy and credibility of information provided by technology-based programs are important aspects that the users are mostly concerned about.

In summary, this study will fill the gap in existing pain management programs for Asian American breast cancer survivors, especially for ABD, and fundamentally enhance the methodology/paradigm related to culturally tailored technology-based programs to reduce health disparities in cancer pain experience among racial/ethnic minority cancer survivors. The design and methods of the program could be easily extended to other sub-ethnic or racial/ethnic groups.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18 years and older who identify as Chinese, Korean, or Japanese;
* have had a breast cancer diagnosis in the past;
* can read and write English, Mandarin (simplified or traditional), Korean, or Japanese;
* have access to the internet through computers or mobile devices (mobile phones and tablets);
* have experienced cancer pain during the past week (at least 1 on a scale from 0 to 5 [no symptom=0, mild symptom that does not bother=1, somewhat bothering symptom=2, moderate symptom=3, severe symptom=4, and worst possible symptom=5]);
* have experienced depressive symptoms during the past two weeks (1 to 10 on the Patient Health Questionnaire) which is equivalent to the cut-point of minimal to moderate depression.

Exclusion Criteria:

* less than 18 years old because their cancer experience would be different from that of adults.
* Those who are in treatment or not in treatment, but who were diagnosed with breast cancer within the past five years, will be excluded.
* Those who participated in the PI's pilot studies will be excluded.
* The participants of R33 phase will exclude those in active depression treatment regardless of their level of depression.
* Those without Internet access will be excluded, but those with Internet access through community/group computers will be included.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Cancer Pain Management (CPM) | Pretest, Post 1-month, Post 3-months
  1 yes/no question on if cancer pain is managed. If yes, additional questions on cancer pain management (types [e.g., acetaminophen, NSAIDs, opioid, massage, acupuncture, acupressure, etc.] and frequency of management & how much relief). If no, what are the reasons.
Brief Pain Inventory-Short Form (BPI-SF) | Pretest, Post 1-month, Post 3-months
  15 items: (a) a global yes or no item asking for a comparison of pain with other minor aches/pains; (b) 4 items (0~10) for the sensory component; (c) 1 item for pain medications; (d) a numerical scale rating the effectiveness of pain relief; (e) 7 items (0~10) for a reactive dimension; and (f) a body diagram for location of pain. The BPI-SF pain scores are determined by adding 4 items on the intensity of pain and 7 items on the interference of pain (0~110; no pain to extreme pain).
Activity monitoring device (Fitbit) as a tool for digital pain biomarkers | Pretest, Post 1-month, Post 3-months
  * Records continuous, automatic, wrist-based resting heart rates, total steps and time (physical activity), and non-walking activities (e.g., swim duration and pool lengths).
  * Has an auto sleep tracking function and records the duration of sleep, sleep stage, and number of times waking. Data on the time asleep and number of wakes will be measured and the time asleep (the overall tracked time - the time awake/restless) will be calculated.
  * The data on resting heart rates, total steps and time (physical activity), and time asleep will be used for data analyses to address the specific aims.
Memorial Symptom Assessment Scale-Short Form (MSAS-SF) | Pretest, Post 1-month, Post 3-months
  * 26 items on symptoms experienced during the past 7 days.
  * Rated on a 5-point (0-4) Likert scale; (0=no symptom to 4=very much).
  * Includes the Global Distress Index (4 psychologic and 6 physical symptoms), the physical symptom distress score (12 items), the psychologic symptom distress score (6 items), the total symptom distress, and the number of total symptoms.
  * Determines the MSAS-SF scores by adding the ratings for distress of 26 symptoms.
Center for Epidemiologic Studies Depression Scale (CES-D) | Pretest, Post 1-month, Post 3-months
  * Measures the frequency of depressive symptoms in the past week.
  * 20 items on the level of depression (range=0~60). All items are summed to calculate depressive symptoms score
Functional Assessment of Cancer Therapy Scale-Breast Cancer (FACT-B) | Pretest, Post 1-month, Post 3-months
  * 44-items to measure multidimensional quality of life in patients with breast cancer.
  * Consists of the FACT-General plus the Breast Cancer Subscale (BCS), which complements the general scale with items specific to quality of life.
  * 7 domains: physical well-being, social/family well-being, emotional well-being, functional well-being, relationship with doctor, BCS, and additional concerns.
  * On a 5-point Likert scale (0=not at all~4=very much), indicating a range of non to extreme interference. All items are summed to obtain a total score (FACT-B score).

SECONDARY OUTCOMES:
Questions on Attitudes and Perceived Barriers | Pretest, Post 1-month, Post 3-months
  6 items on attitudes (bipolar [-3 to +3] scales), 16 items on perceived barriers (4-point Likert scales).
  By summing the items in each subscale, the attitude and perceived barriers scores will be calculated.
Cancer Behavior Inventory (CBI) | Pretest, Post 1-month, Post 3-months
  * A measure of self-efficacy for coping with cancer.
  * 27-items (9-point scale) on how confident to accomplish certain behaviors (not at all=1, to totally confident=9). By summing the items, the self-efficacy scores will be calculated.
Questions on Social Influence | Pretest, Post 1-month, Post 3-months
  Data from 3 items measured on 7-point Likert scales will be summed to calculated the social influence scores.
Disease Factors | Pretest, Post 1-month, Post 3-months
  7 questions on disease factors, including general health, diagnosis of breast cancer, length of time since diagnosis, cancer type (if known), stage of cancer, diagnosed clinical depression and medical treatments, and medication. Used in PSs 1-4, & 5 without any issues.
Genetic factors | Pretest, Post 1-month, Post 3-months
  Questions on family history of depression and psychiatric diseases. 4 questions on family history of depression and other psychiatric diseases only among first-degree relatives (yes or no) and among other relatives (yes or no).
Social Readjustment Rating Scale (SRRS) | Pretest, Post 1-month, Post 3-months
  • 57 items on life events (e.g., death, marriage, empty nest, etc.), giving different weighting depending on the severity of the stressor (0 to 100).
Acculturation Stress Scale (ASS) | pretest, Post 1-month, Post 3-months
  5 questions on the level of acculturation (on a 5-point Likert scale; 1 = exclusively own sub-ethnic group, 5 = exclusively American) in foods, music, customs, close friends, and language (only when the country of birth is not the U.S.).
Personal Resources Questionnaire (PRQ-2000) | pretest, Post 1-month, Post 3-months
  * 15 items measuring perceived level of social support.
  * Includes 7-point Likert scale items in 5 dimensions: (a) provision for attachment/ intimacy; (b) social integration; (c) opportunity for nurturing behavior; (d) reassurance of worth; and (e) the availability of informational, emotional, and material help.
Discrimination Scale (DS) | pretest, Post 1-month, Post 3-months
  • 9 items (6-point Likert scale) on discrimination experience & 1 question on perceived reasons for discrimination 198 (1=ancestor/national origin; 2=gender; 3=race; 4=age; 5=height; 6=skin color; 7=sexual orientation; 8=weight; 9=income or educational level; 10=others).
Perceived Isolation Scale (PIS) | pretest, Post 1-month, Post 3-months
  PIS measures perceived interactions (social isolation) and includes 6 items on social support and 3 items on interactions/loneliness (3-point Likert scales). The average of the items is calculated as the interaction scores.

CONTACTS AND LOCATIONS:
Overall Officials: Eun Ok Im, Principal Investigator — The University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No